CLINICAL TRIAL: NCT05277350
Title: A Phase 1, Randomized, Double-Blind, First-In-Human, Dose Escalation Study Investigating the Safety, Recovery, and Pharmacodynamics of Multiple Oral Administrations of SNIPR001 in Healthy Subjects
Brief Title: A Study Investigating the Safety, Recovery, and Pharmacodynamics of Multiple Oral Administrations of SNIPR001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SNIPR Biome Aps. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: SNIPR001-001
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: E.Coli Infections; Bloodstream Infection
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Dose escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Active Comparator): 6 participants on SNIPR001 (Dose 1 BID for 7 days) and 2 participants on placebo
  Interventions: Drug: SNIPR001; Drug: Placebo
- Cohort 2 (Active Comparator): 6 participants on SNIPR001 (Dose 2 BID for 7 days) and 2 participants on placebo
  Interventions: Drug: SNIPR001; Drug: Placebo
- Cohort 3 (Active Comparator): 12 participants on SNIPR001 (Dose 3 BID for 7 days) and 8 participants on placebo
  Interventions: Drug: SNIPR001; Drug: Placebo

INTERVENTIONS:
Drug: SNIPR001 — SNIPR001 is a live biotherapeutic product consisting of genetically modified bacteriophages specifically targeting Escherichia coli
Drug: Placebo — Matching placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, multiple dose, dose escalation study in healthy participants, investigating the safety, tolerability, recovery, and PD of multiple oral administrations of SNIPR001.

DETAILED DESCRIPTION:
Approximately 36 healthy male and female participants will be randomized to one of 3 active oral doses of SNIPR001 or matching placebo, administered twice a day (BID) for 7 days. Subjects will be followed up until 6 months after receiving the last dose of SNIPR001.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female healthy subject defined as no known clinically relevant organ abnormality, or disease diagnosis, as per Investigator discretion
* No clinically significant abnormalities indicated by safety laboratory test results
* Age between 18 years and 65 years
* E. coli present in feces sample
* Normal defecation pattern (at least once daily)
* Willing to participate in the study and provide fecal samples

Exclusion Criteria:

* Treatment with antibiotics or any other prescription medication within the last 30 days prior to or during screening
* Use of probiotics (not including dairy products) within the last 30 days prior to or during screening
* Smoking (cigarettes, pipes, vaping products, etc.) within the last 3 months prior to or during screening
* 6 months prior to or during screening, recent history of alcohol or drug abuse, or current regular alcohol consumption of more than 14 units per week (one unit of alcohol equals one beer (285 ml), one glass of wine (125 ml), or one glass of spirits (25 ml))
* Positive alcohol or drugs of abuse test
* Pregnancy or lactating or intention of becoming pregnant (all females to agree to use highly effective contraception (defined as those, alone or in combination, that result in a low failure rate i.e., less than 1% per year) for the entire study duration
* Obesity as defined by WHO i.e., BMI>32 kg/m2
* Known to be HIV-positive
* Known active hepatitis B and/or hepatitis C infection
* Known congenital or acquired immunodeficiency
* Allergy to any component of the trial drug and ant-acid treatment
* Regular use of medications that affect gastrointestinal motility e.g., antidiarrheals, stool softeners and laxatives, GLP-1 analogues

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by incidence and severity of AEs and Medically Attended Adverse Events (MAAEs) from the first administration of study drug and up until Day 35 of the study. | 35 days

SECONDARY OUTCOMES:
Incidence and severity of AEs and MAAEs from Day 35 to Day 187 of the study | 152 days
Functional quantification of SNIPR001 (recovery) in feces, blood, and urine before, during, and after multiple oral SNIPR001 administrations | 187 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology, Cincinnati, Ohio, United States